CLINICAL TRIAL: NCT06820931
Title: Indicators and Evaluation of Efficacy of Yin-nourishing and Fire-reducing Chinese Medicine for Girls With Rapid Progression of Early Puberty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: FDCH-ZYXZS-2024313; Z-2019-41-2101-02 (Other Grant/Funding Number: China International Medical Foundation)
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Puberty Changes
Keywords: TCM; puberty

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In this study, 80 patients with premature puberty are included by simple randomization. The randomization scheme is generated by an independent statistical team from the Clinical Trial Center of Children's Hospital of Fudan University using SAS 9.4 software. The intervention protocol determined by the random allocation sequence will be managed by a central coordinator who is not involved in the implementation of the intervention or outcome assessment. The central coordinator will inform the researchers involved in the study of the allocation scheme for the study subjects in accordance with the order in which the guardians of the study subjects sign the informed consent form. The doctor in charge of outcome assessment is completely unaware of the group assignment of the study subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This group does not receive any intervention.
- Intervention group (Experimental): The intervention group is administered drug therapy for a period of six months.
  Interventions: Drug: Xuandi Ziyin Mixture

INTERVENTIONS:
Drug: Xuandi Ziyin Mixture — Treatment is given only with the hospital preparation 'Xuandi Ziyin Mixture' with a dosage of 30ml per administration three times a day.
  Arms: Intervention group

SUMMARY:
1. Evaluate whether AMH and SHBG have differential expression before and after the diagnosis of rapid and slow progression types of early puberty and whether this difference has a predictive effect on the rapid progression type. 2. Assess the therapeutic effect of nourishing yin and purging fire traditional Chinese medicine on girls with rapid progression type of early puberty providing a standardized clinical basis for the formulation of diagnostic and treatment guidelines (or protocols) for the rapid progression type of early puberty using traditional Chinese medicine

ELIGIBILITY:
Inclusion Criteria:

* Girls with an onset age >8 years and ≤9 years;
* Breast bud Tanner stage II breast bud diameter <3 cm;
* Ultrasound examination: unilateral ovarian volume ≥1-3 ml and/or follicle diameter ≥4 mm;
* Bone age does not exceed actual age by more than 1 year;
* LHRH stimulation test: LH/FSH ≥0.6 LH peak ≥5.0 IU/L.
* Good compliance;
* Patients and their parents are willing to actively cooperate with the clinical trial;
* Legal guardian signs the informed consent form.

Exclusion Criteria:

* Disorders of gonadal development such as chromosomal abnormalities hypospadias intersex conditions etc.;
* Use of treatments that affect gonadal function such as chemotherapy radiotherapy;
* Diabetes thyroid dysfunction obesity lipid metabolism disorders or other congenital diseases.

Ages: 8 Years to 9 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The incidence of rapid progression type of precocious puberty | From enrollment to 6 months after treatment.
  The incidence of rapid progression type of precocious puberty between two groups.

SECONDARY OUTCOMES:
AMH | From enrollment to 6 months after treatment.
  Anti-Müllerian Hormone (ng/ml, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
SHBG | From enrollment to 6 months after treatment.
  Sex Hormone Binding Globulin(nmol/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.

OTHER OUTCOMES:
Height | From enrollment to 6 months after treatment.
  The height is measured and obtained by the physician. Place the mechanical height measuring device horizontally on a flat surface, against a wall, and calibrate the height measuring device reading. Instruct the examinee to stand barefoot on the base plate of the height measuring device, facing away from the pillar. When the doctor moves the height measuring device, he holds the handle of the height measuring device, moves horizontally, tries to keep the head upright, and keeps the body and limbs naturally straight. For hair knots and braids that are not convenient to measure height, they should be untied and headwear should be removed. The horizontal pressure plate should be in contact with the head, and the tightness should be moderate. The data is read in cm units and is accurate to 0.1.
Weight | From enrollment to 6 months after treatment.
  The weight is measured and obtained by the physician. Place the electronic scale flat on the ground, calibrate the scale reading, instruct the examinee to empty their bowels and bladder, wear light clothing and stand barefoot naturally in the center of the electronic scale pedal, keep the body stable, record the data, the unit is kg, and the value is accurate to 0.1.
Bone age | From enrollment to 6 months after treatment.
  Bone age is assessed by a radiologist from our hospital through a standard anteroposterior radiograph of the left hand, and is determined according to the Greulich and Pyle (GP) atlas method. The actual age of the child is stated by the parents and then compared by a specialist doctor from our department. Data entry is performed after verification by two individuals.
LH | From enrollment to 6 months after treatment.
  Luteinizing Hormone(U/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
FSH | From enrollment to 6 months after treatment.
  Follicle-Stimulating Hormone(U/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
Estradiol | From enrollment to 6 months after treatment.
  Estradiol(pmol/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
Testosterone | From enrollment to 6 months after treatment.
  Testosterone(nmol/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
PRL | From enrollment to 6 months after treatment.
  Prolactin(mIU/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
Traditional Chinese Medicine syndrome score | From enrollment to 6 months after treatment.
  Traditional Chinese Medicine syndrome score is assessed and obtained by a specialized physician.
  Based on the "Guidelines for the Diagnosis and Treatment of Common Pediatric Diseases in Traditional Chinese Medicine" (Precocious Puberty, ZYYXH/T270-2012) formulated by the China Association of Chinese Medicine and clinical experience, 12 common TCM syndromes for precocious puberty are selected (fear of heat, thirst, facial flushing, "heat in the heart, palms, and soles", preference for fatty and sweet foods, irritability and anger, red and swollen eyes, breast pain, constipation, night sweats, bad breath, red tongue). Each item is worth 2 points, with 2 points for presence, 1 point for improvement, and 0 points for absence. The syndrome score is obtained by adding them together.
Breast Tanner staging | From enrollment to 6 months after treatment.
  Breast Tanner staging (obtained by the physician through physical examination). The Tanner staging criteria and standard illustrations are used for definition. Some obese girls may find it difficult to distinguish between breast tissue and fat tissue, so we have all the subjects raise their arms and have professional doctors use visual and palpation methods to assess the breast development stage.
Uterine volume | From enrollment to 6 months after treatment.
  Uterine volume obtained through ultrasound measurement; The size and shape of the organs are measured by a professional ultrasound physician from our hospital. The volume is calculated using the formula: V=(π /6)*length*anteroposterior diameter*transverse diameter, with the unit being cubic centimeters (cm³).
ovarian volume | From enrollment to 6 months after treatment.
  Ovarian volume obtained through ultrasound measurement The size and shape of the organs are measured by a professional ultrasound physician from our hospital. The volume is calculated using the formula: V=(π /6)*length*anteroposterior diameter*transverse diameter, with the unit being cubic centimeters (cm³).
follicle diameter | From enrollment to 6 months after treatment.
  Follicle diameter obtained through ultrasound measurement The size and shape of the organs are measured by a professional ultrasound physician from our hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided